CLINICAL TRIAL: NCT03945760
Title: An Investigator Initiated Study to Evaluate the Efficacy of Baricitinib In Treatment of Delayed-Type Hypersensitivity Versus Irritant Skin Reactions In Healthy Adult Male Subjects
Brief Title: Efficacy of Baricitinib In Treatment of Delayed-Type Hypersensitivity Versus Irritant Skin Reactions in Healthy Adult Male Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wright State Physicians (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: I4V-US-O007
Record Dates: First submitted 2019-04-26; First posted 2019-05-10 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Allergic Contact Dermatitis
MeSH Terms: conditions — Dermatitis, Allergic Contact | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Subjects Taking Baricitinib 2 mg (Experimental): Subjects will be taking Baricitinib 2mg
  Interventions: Drug: Baricitinib
- Subjects Taking Placebo (Placebo Comparator): Subjects will be taking placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Baricitinib 2 mg
  Arms: Subjects Taking Baricitinib 2 mg
Drug: Placebo — Placebo
  Arms: Subjects Taking Placebo

SUMMARY:
The treatment of allergic contact dermatitis (ACD) can be unsatisfactory, and that other skin diseases such as atopic dermatitis have an increased likelihood of ACD, improved systemic treatments are needed.

This research study explores the effectiveness of Baricitinib in treating Delayed-Type Hypersensitivity (allergic) versus Irritant Skin reactions. Subjects for this study need to be healthy males between the ages of 18 and 40. This study will evaluate this by injecting antigens as well as applying them on top of the skin to the forearm then measure the effects of Baricitinib by skin and blood testing.

ELIGIBILITY:
Inclusion Criteria:

* Males 18-40 years of age at the time of signing the informed consent document
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted
* Able to adhere to the study visit schedule and other protocol requirements
* Must be in good health as judged by the Investigator, based on medical history and physical examination, and no laboratory abnormalities

Exclusion Criteria:

* Any known severe allergies to yeast products
* Currently active skin diseases such as psoriasis, atopic dermatitis, allergic contact dermatitis or irritant contact dermatitis
* Inability to understand informed consent
* Any medical condition that the investigator feels would interfere with study
* Any abnormalities on physical exam or screening laboratory studies (to progress to Part II)
* Agree to discontinue use of prohibited medications at least 4 weeks prior to screening:

topical corticosteroids, oral or injectable systemic steroids, systemic immunomodulators (cyclosporine, methotrexate, etc.), oral or topical antihistamines

* Positive reaction to tuberculin test (PPD) or negative control
* Negative reaction to initial skin testing for Candida, Trichophyton, or Sodium Laurel Sulfate

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with reduced skin inflammation associated with Delayed-Type Hypersensitivity (DTH) versus irritant skin reactions by erythema measurement. | Day 28
  Investigator will assess the skin inflammation reduction as measured by erythema associated with DTH versus irritant skin reactions.
Number of participants with reduced skin inflammation associated with Delayed-Type Hypersensitivity (DTH) versus irritant skin reactions by measurement of reaction size. | Day 28
  Investigator will assess the skin inflammation reduction as measured by reaction size associated with DTH versus irritant skin reactions.
Number of participants with reduced skin inflammation associated with Delayed-Type Hypersensitivity (DTH) versus irritant skin reactions by pro-inflammatory cytokine profile. | Day 28
  Investigator will assess the skin inflammation reduction as measured by pro-inflammatory cytokine profile associated with DTH versus irritant skin reactions.

SECONDARY OUTCOMES:
Number of participants with reduced pruritus associated with DTH versus irritant skin reactions. | Day 28
  Investigator will assess pruritus reduction associated with DTH versus irritant skin reactions by a daily itch rating scale questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Travers, MD, PhD, Principal Investigator — Wright State Physicians
Locations (1):
- Wright State Physicians, Fairborn, Ohio, United States